CLINICAL TRIAL: NCT00785356
Title: A Multi-Center, Placebo Controlled, Safety and Efficacy Study of the Selective Progesterone Receptor Modulator Proellex® (CDB-4124) in Anemic, Pre-Menopausal Women With Symptomatic Uterine Fibroids Requiring Hysterectomy
Brief Title: Safety and Efficacy of Proellex in Pre-Menopausal Anemic Women With Symptomatic Uterine Fibroids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Repros stopped the study for safety and FDA put the study on hold for safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZPU-302
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids; Anemia
Keywords: Uterine fibroids; Anemia
MeSH Terms: conditions — Leiomyoma; Anemia | interventions — telapristone acetate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 25 mg Proellex (Experimental): Proellex 25 mg
  Interventions: Drug: Proellex 25 mg
- Proellex 50 mg (Experimental): Proellex 50 mg
  Interventions: Drug: Proellex 50 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proellex 25 mg — Proellex 25 mg, 1 - 25 mg capsule and 1 placebo capsule daily for 3 months
  Other Names: Telapristone acetate
  Arms: 25 mg Proellex
Drug: Proellex 50 mg — Proellex 50 mg, 2 - 25 mg capsules daily for 3 months
  Other Names: Telapristone acetate
  Arms: Proellex 50 mg
Drug: Placebo — Placebo, 2 capsules daily for 3 months
  Other Names: Sugar pill; Dummy
  Arms: Placebo

SUMMARY:
Subjects will be randomly assigned to one of 3 treatment groups and receive 325 mg (65 mg elemental iron) iron supplements twice daily.

DETAILED DESCRIPTION:
Eligible female subjects will be randomly assigned to one of the three treatment groups. Subjects will receive 325 mg (65 mg elemental iron) iron supplements to be taken twice daily during study drug treatment. The study duration is approximately six months, which is comprised of a 4 - 6 week screening period, a three-month drug treatment period, and a one-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Female, between the ages of 18 and 48 years with Body Mass Index (BMI) between 18 and 39, inclusive;
* Anemic, defined as hemoglobin levels less than or equal to 10.5 g/dL and uterine fibroid-associated symptoms indicated by a history of excessive menstrual bleeding;
* Surgical interventions for uterine fibroids (e.g. hysterectomy or myomectomy) planned or anticipated after the study;
* Willing to comply with all study procedures, including the endometrial biopsies and blood draws for all visits, including Follow-up Visits

Exclusion Criteria:

* Post-menopausal women or women likely to become post-menopausal during the study, defined as one or more of the following:

  * Six months or more (immediately prior to Screening Visit) without a menstrual period, or
  * Prior hysterectomy, or
  * Prior bilateral oophorectomy (unilateral oophorectomy is not exclusionary if regular menstruation is occurring);
* Females who have undergone a uterine arterial embolization, or endometrial ablation therapy (previous myomectomy is acceptable) for any cause;
* Documented endometriosis or active pelvic inflammatory disease (PID);
* Having a diagnosis, or suspected diagnosis, of carcinoma of the breast or reproductive organs;
* Known active infection with HIV, Hepatitis A, B or C, Gonorrhea, or Chlamydia;
* Use of prohibited concomitant medications:

  1. Depo-Provera use must cease ten months prior to first dose of study drug, or
  2. GnRH agonists use (e.g. Lupron Depot) must cease six months prior to first dose of study drug, or
  3. Oral contraceptive or other hormonal treatments use must cease for 30 days prior to the start of the study

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (7):
- Mexico (7):
  - Hospital Perinatal del Estado de Mexico del ISEM, Toluca, Estado de Mexico C.P.
  - Comité para la Prevención de la Osteoporosis COMOP, Mexico City, Federal District
  - Centro Hospitalario Nuevo Sanatorio Durango, Mexico City, Federal District
  - Instituto Nacional de Perinatología "Isidro Espinosa de los Reyes", Mexico City, Federal District
  - Hospital de la Fe, San Miguel de Allende, Guanajuato
  - Hospital Universitario "Dr. José Eleuterio González" Facultad de Medicina de la Universidad Autónoma de Nuevo León (UANL), Monterrey, Nuevo León
  - MIRC (Monterrey International Research Center), Monterrey, Nuevo León

RESULTS

PARTICIPANT FLOW:
Groups:
- All Groups: Proellex 25 mg, Proellex 50 mg, 1placebo
Period: Overall Study
Arm/Group | All Groups
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study prematurely terminated | 8

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg Proellex | Proellex 50 mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Comparison Between the 50 mg Proellex® Dose Level and Placebo in the Change in Hemoglobin From Baseline to 3 Months.
Time Frame: 3 months
Arm/Group | 25 mg Proellex | Proellex 50 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: No adverse events data is available.
Arm/Group | 25 mg Proellex | Proellex 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights